CLINICAL TRIAL: NCT06016322
Title: The Effect of Dried Chicory Root on Inflammation, Gut Microbiota and Complaints in Patients With Inflammatory Bowel Disease: a Pilot Study
Brief Title: Dried Chicory Root in IBD
Acronym: Chic-IBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: WholeFiber (Unknown); MyMicroZoo (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NL85061.042.23; KIEM.K23.01.148 (Other Grant/Funding Number: NWO)
Record Dates: First submitted 2023-08-08; First posted 2023-08-29 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Inflammatory Bowel Diseases; Dietary Exposure
Keywords: Inflammatory bowel disease; dietary fiber; gut microbiome; inflammation
MeSH Terms: conditions — Inflammatory Bowel Diseases; Inflammation

STUDY DESIGN:
Intervention Model Description: Pilot study investigating the effect of additional dietary intake 10-20 gram of a dried vegetable fibre. The difference in outcomes before and after the intervention in fecal calprotectin, IBD complaints, QOL, serum inflammatory markers, gut microbiota and SCFA will be determined
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Before and after study in 6 patients with UC and 6 patients wiht CD (Experimental): This is a 4-week before-after pilot study to explore the effectiveness of a WholeFiber Trademark (TM) intervention (a dried vegetable rich in prebiotic intrinsic fibers) on inflammation, fecal gut microbiota and metabolites, IBD-complaints and QoL and assesses its feasibility. In this before-after study, 12 patients with IBD will receive WholeFiberTM; of which 6 patients with CD and 6 patients with UC to assess if there is a difference in effect between these groups of patients.
  Interventions: Dietary Supplement: Dried Chicory Root

INTERVENTIONS:
Dietary Supplement: Dried Chicory Root — Subjects will receive 1 sachet of 10g WholeFiberTM for the first 2 weeks (equals 8.5 g fiber), and 2 sachets of 10g WholeFiberTM per day for the last two weeks (equals 17 g fiber).
  WholeFiberTM is a fiber-rich dried vegetable made from the chicory root that contains four types of prebiotic fibers (inulin, pectin, cellulose, hemi-cellulose).
  Other Names: WholeFiber Trademark (TM)

SUMMARY:
The goal of this clinical pilot trial is to test the use of dried chicory root in patients with IBD. The main questions it aims to answer are:

what the effect of a 4-week 10-20 g/day WholeFiberTM intervention on fecal calprotectin, IBD-complaints and QoL, serum inflammatory markers, gut microbiota and SCFA levels in patients with Crohn's disease and ulcerative colitis Participants will receive 1 sachet of 10g WholeFiberTM for the first 2 weeks (equals 8.5 g fiber), and 2 sachets of 10g WholeFiberTM per day for the last two weeks (equals 17 g fiber).

Researchers will compare the above mentioned outcomes before and after the intervention.

DETAILED DESCRIPTION:
Rationale: Inflammatory Bowel Diseases (IBD), of which Ulcerative Colitis (UC) and Crohn's Disease (CD) are the main types, includes recurring episodes of inflammation in the gastro-intestinal tract and severely impacts quality of life (QoL), leads to more hospitalization and increases the mortality risk. An impaired gut microbiota and lower levels of short-chain fatty acids (SCFA) have been linked to the pathophysiology. A higher fiber intake is linked to positive changes in the gut microbiota and increase SCFA-production, however patients with IBD consume too little dietary fiber. WholeFiberTM, a dried vegetable rich in 4 types of prebiotic fiber, may be an easy solution to increase dietary fiber intake, impact the gut microbiota and SCFA, IBD-complaints and health parameters.

Objective: To explore the effect of a 4-week 10-20 g/day WholeFiberTM intervention on fecal calprotectin, IBD-complaints and QoL, serum inflammatory markers, gut microbiota and SCFA levels in patients with CD and UC.

Study design: this is a 4-week pilot study with one arm to explore the effects of a WholeFiberTM intervention. Measurements will take place before and after the intervention, questionnaires will also be conducted halfway.

Study population: in total 12 patients with mild to moderate IBD complaints will be included, of which 6 UC and 6 CD patients, to investigate if there is a difference between the two groups in efficacy of WholeFiberTM.

Intervention: Subjects will receive 1 sachet of 10g WholeFiberTM for the first 2 weeks (equals 8.5 g fiber), and 2 sachets of 10g WholeFiberTM per day for the last two weeks (equals 17 g fiber).

Main study parameters/endpoints: the primary parameter is change in fecal calprotectin after the 4-week intervention, which is a marker for inflammation in the gut. Secondary parameters are improvements in IBD-complaints, QoL, serum markers, and changes in the gut microbiota and increase in fecal SCFA-production. Moreover, it will be explored whether the response on the intervention will be different between UC and CD. Furthermore, an evaluation questionnaire will be conducted to assess feasibility and acceptance of the WholeFiberTM intervention in this population.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥18 years;
* Having a diagnosis of IBD (either UC or CD) and undergoing treatment at the policlinic at the University Medical Center Groningen;
* Mild or moderate IBD, defined as fecal calprotectin levels ≥100 μg and Harvey Bradshaw Index (HBI) <8 for CD patients or Simple Clinical Colitis Activity Index (SCCAI) <5 for UC patients;
* Using stable maintenance therapy for at least 12 weeks;
* Being able to read and speak Dutch;
* Willing to come to the University Medical Center Groningen for practical reasons (visiting the study site);
* Willing to continue their regular lifestyle patterns during the study.

Exclusion Criteria:

* Having a medical history that may impact study outcomes, such as a diagnosis of diabetes mellitus type 2, heart disease, renal disease, cancer, celiac disease;
* Having an ileostomy or colostomy, as this greatly impacts bowel function and gut microbiota composition;
* Having a clinically significant stenosis;
* Use of antibiotics <4 weeks before study start;
* Use of prebiotics, probiotics and/or synbiotic (this should be stopped 4 weeks before start of the study) or other fiber supplements such as psyllium;
* Use of tube feeding or sib-feeding;
* Being pregnant or lactating;
* Participation in another clinical study at the same time;
* Unable or unwilling to comply to study rules

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-10-02 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
change in fecal calprotectin | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week 10-20 g/day WholeFiberTM intervention on fecal calprotectin levels in patients with CD and UC.

SECONDARY OUTCOMES:
Change in IBD complaints by HBI for CD | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention on IBD-complaints in patients with CD measured by the Harvey Bradshaw Index (HBI)
Change in IBD complaints by SCCAI for UC | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention on IBD-complaints in patients UC measured by the Simple Clinical Colitis Activity Index (SCCAI)
Change in QOL measured by IBDQ | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on QoL measured by the IBDQ (Irvine 1999)
Change in the Food-related Quality of Life (FrQOL) | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on Food-related QoL measured by a validated instrument by Hughes et al 2015
Change in stool consistency | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on stool consistency. Stool consistency will be measured using the validated Bristol Stool Chart.
Change in stool frequency | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on stool frequency. Patients will be asked how often they defecated per day during the past week
Change in fecal microbiota composition: Shannon-index | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on fecal microbiota composition. Next generation sequencing will be used ot determine bacterial richness (Shannon-index)
Change in fecal microbiota composition by beta-diversity | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on fecal microbiota composition. Next generation sequencing will be used ot determine bacterial interindividual variations (beta-diversity)
Change in fecal SCFA levels: lactate | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention on fecal lactate in patients with CD and UC measured by a conductivity detector.
Change in fecal SCFA levels: formate | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention on fecal formate in patients with CD and UC measured by a conductivity detector.
Change in fecal SCFA levels; butyrate | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention on fecal butyrate in patients with CD and UC measured by a conductivity detector.
Change in fecal SCFA levels: propionate | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention on fecal propionate in patients with CD and UC measured by a conductivity detector.
Change in fecal SCFA levels: acetate | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention on fecal acetate in patients with CD and UC measured by a conductivity detector.
Change in fecal acidity (pH) | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on fecal acidity (pH) by a PCE-228-R pH and redox meter in a stool sample.
Change in fecal redox status | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on fecal redox status, measured by PCE-228-R instrument.
Change in serum leukocytes | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on leukocytes count.
Change in serum thrombocytes | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on thrombocytes.
Change in serum iron status: serum iron | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC serum iron [micromol/L]
Change in serum iron status: Total Iron Binding Capacity (TIBC) | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on Total Iron Binding Capacity (TIBC) [micromol/L]
Change in serum iron status: ferritin | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on ferritin [microg/L]
Change in serum iron status: transferrin | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on transferrin [g/L]
Change in serum ALAT | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on Alanine Aminotransferase (ALAT).
Change in serum ASAT | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on Aspartate Aminotransferase (ALAT).
Change in serum GGT | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on Gamma-Glutamyl Transferase (GGT)
Change in serum creatinine | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on iron status.
Change in C-reactive protein (CRP) | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on C-reactive protein (CRP), which is an inflammation marker.
Change in inflammatory marker IL-6 analysed by an ELISA kit | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on the inflammatory marker IL-6 on an ELISA kit
Change in inflammatory marker IL-8 analysed by an ELISA kit | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on the inflammatory marker IL-8 on an ELISA kit
Change in inflammatory marker IL-10 analysed by an ELISA kit | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on the inflammatory marker IL-10 on an ELISA kit
Change in inflammatory markers IL-12 analysed by an ELISA kit | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on the inflammatory marker IL-12 on an ELISA kit
Change in inflammatory markerIL-17a analysed by an ELISA kit | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on the inflammatory marker IL-17a on an ELISA kit
Change in inflammatory marker IL-22 analysed by an ELISA kit | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on the inflammatory marker IL-22 on an ELISA kit
Change in inflammatory marker IL-23 analysed by an ELISA kit | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on the inflammatory marker IL-23 on an ELISA kit
Change in inflammatory marker TNF-alpha analysed by an ELISA kit | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on the inflammatory marker TNF-alpha on an ELISA kit
Change in inflammatory marker Interferon(IFN)-gamma analysed by an ELISA kit | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on the inflammatory marker Interferon(IFN)-gamma on an ELISA kit
Change in oxidative stress measured by free thiols | difference between baseline and after 4-week intervention
  To explore the effect of a 4-week WholeFiberTM intervention in patients with CD and UC on oxidative stress measured by free thiols.

OTHER OUTCOMES:
Difference in change in fecal calprotectin between patients with CD and UC | difference between baseline and after 4-week intervention
  To explore the difference between CD an UC in change in the effect of a 4-week 10-20 g/day WholeFiberTM intervention on fecal calprotectin levels
Appreciation of WholeFiberTM evaluated by patients with CD and UC? | after 4-week intervention
  How participants with CD and UC appreciated of WholeFiberTM by chosing a digit on a vascale from 1 to 10, being 1 the lowest number of appreciation and 10 the highest number
The convenience of the use of WholeFiberTM evaluated by patients with CD and UC? | after 4-week intervention
  Participants are asked to rate the following statement "I find Whole Fiber easy to use" and can answer on a Lickert with 5 different categories: 1. completely disagree 2. disagree 3. neutral, 4 agree 5. completely agree.
The palatability of the use of WholeFiberTM evaluated by patients with CD and UC? | after 4-week intervention
  Participants are asked to rate the following statement "I find Whole Fiber tasty to eat" and can answer on a Lickert with 5 different categories: 1. completely disagree 2. disagree 3. neutral, 4 agree 5. completely agree.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Puhlmann ML, de Vos WM. Back to the Roots: Revisiting the Use of the Fiber-Rich Cichorium intybusL. Taproots. Adv Nutr. 2020 Jul 1;11(4):878-889. doi: 10.1093/advances/nmaa025. PMID 32199025
- [Result] Peters V, Dijkstra G, Campmans-Kuijpers MJE. Are all dietary fibers equal for patients with inflammatory bowel disease? A systematic review of randomized controlled trials. Nutr Rev. 2022 Apr 8;80(5):1179-1193. doi: 10.1093/nutrit/nuab062. PMID 34486663
- [Result] Puhlmann ML, de Vos WM. Intrinsic dietary fibers and the gut microbiome: Rediscovering the benefits of the plant cell matrix for human health. Front Immunol. 2022 Aug 18;13:954845. doi: 10.3389/fimmu.2022.954845. eCollection 2022. PMID 36059540
- See also: Dried Chicory Root Improves Bowel Function, Benefits Intestinal Microbial Trophic Chains and Increases Faecal and Circulating Short Chain Fatty Acids in Subjects at Risk for Type 2 Diabetes — https://www.cambridge.org/core/journals/gut-microbiome/article/dried-chicory-root-improves-bowel-function-benefits-intestinal-microbial-trophic-chains-and-increases-faecal-and-circulating-short-chain-fatty-acids-in-subjects-at-risk-for-type-2-diabetes/6209AEAFBDDB181197F22AE24388186B